CLINICAL TRIAL: NCT03538288
Title: A Pilot Trial Determining the Feasibility of Delivering Twenty Treatments of Repetitive Transcranial Magnetic Stimulation (rTMS) to Treatment Seeking Cannabis Use Disordered Participants
Brief Title: Feasibility Trial of rTMS for Cannabis Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00054706
Record Dates: First submitted 2016-09-07; First posted 2018-05-29 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-05

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Twenty sessions of rTMS (Experimental): Twenty sessions of rTMS will be applied to treatment seeking participants.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — rTMS will be applied at 10 Hz to the DLPFC

SUMMARY:
This small pilot trial will recruit 10 cannabis use disordered participants and apply 20 sessions of rTMS in conjunction with a two session Brief Marijuana Dependance Counseling treatment paradigm. The investigators are primarily seeking to determine if the proposed paradigm is feasible and well tolerated.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to investigate if a course of excitatory DLPFC rTMS is feasible and well tolerated by a group of treatment seeking CUD patients (Aim1). The investigators are also hoping to preliminarily determine if a course of rTMS reduces cannabis cue-induced craving (Aim2). Additionally the investigators want to preliminarily explore the mechanistic underpinnings of any observed effect by collecting functional magnetic resonance imaging (fMRI) data during cannabis cue-administration before and after the treatment course (Aim 3). These aims will be addressed through an open label study in which 10 treatment seeking cannabis use disordered participants will be given 20 sessions of Active excitatory rTMS applied to the DLPFC. TMS will be delivered in an accelerated fashion over two weeks (2 sessions each day, five days each week). TMS will be applied in conjunction with a validated two-session Motivational Enhancement Therapy (MET) behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Participants must be between the ages of 18 and 60.
3. Participants must meet DSM-5 criteria for at least moderate Cannabis Use Disorder, with use of at least 20 / last 28 days.
4. Participants must express a desire to quit cannabis.
5. Participants must have a positive UDS for cannabis during their enrollment visit (confirming they are regular users).

Exclusion Criteria:

1. Participants must not be pregnant or breastfeeding.
2. Participants must not test positive for any substance other than cannabis on UDS during their enrollment visit.
3. Participants must not meet moderate or severe use disorder of any other substance with the exception of Tobacco Use Disorder.
4. Participants must not be on any medications that have central nervous system effects.
5. Participants must not have a history of/or current psychotic disorder or bipolar disorder.
6. Participants must not have any other Axis I condition requiring current treatment and must have a HRSD24 ≤10 indicating no clinically relevant depressive symptoms.
7. Participants must not have a history of dementia or other cognitive impairment.
8. Participants must not have active suicidal ideation or a suicide attempt within the past 90 days.
9. Participants must not have any contraindications to receiving rTMS (e.g. metal implanted above the head, history of seizure, any known brain lesion).
10. Participants must not have any unstable general medical conditions.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Determine if a course of rTMS is feasible to deliver and well tolerated by a group of cannabis use disordered participants. | 7 weeks
  The investigators will test the hypothesis that at least 50% of enrolled participants will complete the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, Principal Investigator — Instructor
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided